CLINICAL TRIAL: NCT00920179
Title: The Application of In Vivo Confocal Scanning Laser Microscopy in the Evaluation of the Secretory Glands in Patients With Sjögren's Syndrome
Brief Title: Confocal Microscopy and Lacrimal Gland in Sjogren's Syndrome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Keio University (Other)
Responsible Party: Associate Professor Dr Murat Dogru, J&J Ocular Surface and Visual Optics Department
Other Study IDs: 21071965
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Primary Sjogren's Syndrome
Keywords: dry eye, in vivo confocal microscopy, inflammation, acinar unit density, lacrimal gland
MeSH Terms: conditions — Dry Eye Syndromes; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dry eye group: Dry eye patients with Primary Sjogren's syndrome
- Controls: Healthy subjects without dry eyes

SUMMARY:
Traditional methodological clinical and instrumental diagnostics of the lacrimal gland for the study of glandular architecture and functions are limited and include analysis of tear constituents, evaluation of apparent diffusion coefficients in magnetic resonance imaging and histopathological evaluation of lacrimal gland biopsy specimens. Confocal microscopy is a new emerging technology which is useful as a supplementary diagnostic tool for in vivo assessment of anterior-segment disorders.The use of in vivo confocal microscopy in a comparative study of the microscopic morphology of the salivary/lacrimal glands have not been reported up to date. In this study, we employ laser scanning confocal microscopy to evaluate the morphological changes of the salivary/lacrimal glands in patients with primary Sjögren's syndrome and compare the results with those of healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* The Sjögren's syndrome diagnosis was made according to the revised American-European consensus criteria.
* Briefly, the patients had to have ocular and oral symptoms of dryness,
* clinically diagnosed dry eye and dry mouth disease,
* serum rheumatoid factor and antinuclear antibody levels ≥1:160,
* positive serology for anti SS-A or anti SS-B antibodies,
* labial salivary gland inflammatory infiltration focus score ≥2 and consents for lacrimal gland biopsy to be included into this study.

Exclusion Criteria:

* Patients with any history of ocular surgery including punctal occlusion,
* other ocular or systemic disease
* or a history of topical/ systemic drug use or contact lens wear or
* other systemic disorders that would cause dry eyes or that would alter the ocular surface.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary SS and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cell density | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Tsubota, Professor, Study Director — Keio University
Locations (1):
- Keio University School of Medicine, Tokyo, Japan